CLINICAL TRIAL: NCT04875299
Title: Evaluation of the Optimal Concentration Range of Adalimumab for Ankylosing Spondylitis in a Prospective Observational Study
Brief Title: Optimal Adalimumab Plasma Concentrations in Ankylosing Spondylitis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine (Other); Central South University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Tianjin First Central Hospital (Other); Wuxi No. 2 People's Hospital (Other); The First People's Hospital of Changzhou (Other); Affiliated Hospital of Nantong University (Other); Shandong Provincial Hospital (Other Government); Qingdao Municipal Hospital (Other); Liaocheng People's Hospital (Other); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Miao Liyan, vice president, The First Affiliated Hospital of Soochow University
Other Study IDs: ADL-TDM-02
Record Dates: First submitted 2021-04-29; First posted 2021-05-06 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; adalimumab
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma and DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- adalimumab TDM: Patients with active ankylosing spondylitis receiving adalimumab treatment.
  Interventions: Other: The study is observational

INTERVENTIONS:
Other: The study is observational — The study is observational

SUMMARY:
The optimal plasma concentration range of adalimumab in Chinese patients with active ankylosing spondylitis remains unknown, the aims of this study is to determine the concentration-effect relationship, and explore the effect of anti-drug antibody or biomarkers on clinical outcomes in a real-world setting.

DETAILED DESCRIPTION:
This prospective observational study will include Chinese adult patients with active ankylosing spondylitis receiving adalimumab treatment. The primary outcome is the mean change from baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS).

ELIGIBILITY:
Inclusion Criteria:

1. Consent of the patient.
2. Patient who meets the definition of Ankylosing Spondylitis based on the 1984 Modified New York Criteria, has a diagnosis of active Ankylosing Spondylitis (BASDAI ≥ 4, Back pain ≥ 4).
3. Patients who have indication of adalimumab.
4. Patients on NSAIDs treatment need to be on a stable dose for at least 4 weeks.

Exclusion Criteria:

(1) Hepatitis B or tuberculosis patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective observational study will include Chinese adult patients with active ankylosing spondylitis receiving adalimumab treatment.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in ASDAS | Week 24
  ASDAS will be measured at week 24 and will be compared to baseline

SECONDARY OUTCOMES:
ASAS20 response | Week 2, 4, 8, 12, 24
  ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) subjects. ASAS has 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 20 = 20% improvement (vs. baseline) and an absolute improvement ≥ 10 units on a 0-100 scale (0 = no disease activity; 100 = high disease activity) for ≥ 3 domains, and no worsening (defined as a worsening of ≥ 20% and a net worsening of ≥ 10 units) in the remaining domain.
ASAS40 response | Week 2, 4, 8, 12, 24
  ASAS 40 = 40% improvement (vs. baseline) and an absolute improvement ≥ 20 units on a 0-100 scale (0 = no disease activity; 100 = high disease activity) for ≥ 3 domains, and no worsening (defined as a worsening of ≥ 20% and a net worsening of ≥ 10 units) in the remaining domain.
BASDAI50 response | Week 2, 4, 8, 12, 24
  Utilizing a Visual Analog Scale (VAS) of 0-10 (0=none and 10=very severe) subjects answered 6 questions measuring discomfort, pain, fatigue, and morning stiffness. BASDAI 50 = at least 50% improvement (vs. baseline) in BASDAI.
ASDAS response | Week 2, 4, 8, 12, 24
  A decrease in ASDAS from baseline (△ASDAS) ≥ 2.0 or a moderate disease activity achievement (ASDAS < 2.1) with △ASDAS ≥ 1.1 is considered as response
ASDAS remission | Week 2, 4, 8, 12, 24
  ASDAS < 2.1 at assessment time point is considered as remission
Safety analysis - Occurence of adverse event | Week 24
  Safety analysis include occurence of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Ph.D, Study Chair — The Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No